CLINICAL TRIAL: NCT03409744
Title: An Open-Label Study to Evaluate the Long-Term Safety and Efficacy of Evinacumab in Patients With Homozygous Familial Hypercholesterolemia
Brief Title: Evaluate the Long-Term Safety and Efficacy of Evinacumab in Patients With Homozygous Familial Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R1500-CL-1719; 2017-003170-13 (EudraCT Number)
Record Dates: First submitted 2018-01-08; First posted 2018-01-24 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Homozygous Familial Hypercholesterolemia
Keywords: HoFH
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — evinacumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- evinacumab (Experimental)
  Interventions: Drug: evinacumab

INTERVENTIONS:
Drug: evinacumab — Intravenous (IV) administration
  Other Names: REGN1500; EVKEEZA®

SUMMARY:
The primary objectives of the study are:

* To evaluate the long-term safety and tolerability of evinacumab in patients with Homozygous Familial Hypercholesterolemia (HoFH)
* To evaluate the long-term safety and tolerability of evinacumab in adolescent patients with HoFH

The secondary objectives of the study are:

* To evaluate the effect of evinacumab on lipid parameters in patients with HoFH
* To evaluate the effect of evinacumab on lipid parameters in adolescent patients with HoFH
* To evaluate the potential development of anti-evinacumab antibodies

ELIGIBILITY:
Key Inclusion Criteria:

1. Completion of the parent study in which they participated
2. Able to understand and complete study-related questionnaires

Key Exclusion Criteria:

1. Significant protocol deviation in the parent study based on the investigator's judgment, such as non-compliance by the patient
2. Concomitant medications that have not been stable prior to the baseline visit
3. Adverse event leading to permanent discontinuation from parent study
4. Any new condition or worsening of an existing condition, which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study
5. Member of the clinical site study team and/or his/her immediate family
6. Pregnant or breastfeeding women
7. Women of childbearing potential who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 24 weeks after the last dose of study drug
8. Men who are sexually active with women of childbearing potential and are unwilling to use the following forms of medically acceptable birth control during the study drug treatment period and for 24 weeks after the last injection of study drug: vasectomy with medical assessment of surgical success OR consistent use of a condom.

Note: Other protocol defined Inclusion/Exclusion criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (36):
- United States (8):
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Boca Raton, Florida
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Cincinnati, Ohio
  - Clinical Trial Site, Portland, Oregon
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Dallas, Texas
- Australia (2):
  - Clinical Trial Site, Camperdown, New South Wales
  - Clinical Trial Site, Perth, Western Australia
- Austria (2):
  - Regeneron Study Site, Vienna, Vienna
  - Regeneron Study Site, Innsbruck
- Canada (2):
  - Clinical Trial Site, Chicoutimi, Quebec
  - Clinical Trial Site, Québec
- Regeneron Study Site, Prague, Kateřinská, Czechia
- France (3):
  - Clinical Trial Site, Paris, Cedex 13
  - Clinical Trial Site, Marseille, Cedex 5
  - Clinical Trial Site, Dijon, Cedex
- Greece (2):
  - Regeneron Study Site, Kallithea, Athens
  - Clinical Trial Site, Ioannina
- Italy (2):
  - Clinical Trial Site, Napoli, Campania
  - Clinical Trial Site, Roma, Rome
- Japan (6):
  - Clinical Trial Site, Ōbu, Aichi-ken
  - Regeneron Study Site, Kurume, Fukuoka
  - Regeneron Study Site, Nishinomiya, Hyōgo
  - Regeneron Study Site, Kanazawa, Ishikawa-ken
  - Regeneron Study Site, Kita-ku, Osaka
  - Regeneron Study Site, Suita, Osaka
- Clinical Trial Site, Amsterdam, Netherlands
- South Africa (2):
  - Regeneron Study Site, Johannesburg, Gauteng
  - Regeneron Study Site, Cape Town, Western Cape
- Ukraine (5):
  - Clinical Trial Site, Ivano-Frankivsk
  - Clinical Trial Site #1, Kharkiv
  - Clinical Trial Site #2, Kharkiv
  - Clinical Trial Site, Kyiv
  - Rgeneron Study Site, Kyiv

REFERENCES:
- See also: A Plain Language Summary is available on TrialSummaries.com — https://www.trialsummaries.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 118 participants were planned to be enrolled. 116 participants were enrolled & treated. Reasons for screen fail were: 1 participant was unwilling to use protocol defined contraception, and 1 participant had a Low-density lipoprotein cholesterol (LDL-C) level less than the lower limit required for inclusion.
Groups:
- Total Evinacumab: Includes all participants who were enrolled and received at least 1 dose or part of a dose of open-label study treatment.
Period: Overall Study
Arm/Group | Total Evinacumab
Started | 116
Completed | 106
Not Completed | 10
Not completed — Death | 2
Not completed — Physician Decision | 5
Not completed — Pregnancy | 1
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Total Evinacumab
Number analyzed (Participants) | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.8 (15.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 80
  Black or African American | 4
  Asian | 12
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0
  Not Reported | 11
  Other | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Up to Week 216
Description: The safety analysis set (SAF) included all participants who were enrolled and received at least 1 dose or part of a dose of open-label study treatment.
Time Frame: Up to 216 weeks
Measure: Number; unit: Number of participants
Groups:
- Overall Study Total Evinacumab: Includes all participants who were enrolled and received at least 1 dose or part of a dose of open-label study treatment.
Arm/Group | Overall Study Total Evinacumab
Number analyzed (Participants) | 116
Number of participants
  Participants with any TEAE | 93
  Participants with at least one serious TEAE | 27

2. Secondary Outcome: Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) Over Time
Description: as for outcome 1
Time Frame: Up to 120 weeks
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Overall Study Total Evinacumab
Number analyzed (Participants) | 116
Percentage of change
  Week 8: number analyzed (Participants) | 109
  Week 8 | -46.45 (35.504)
  Week 24: number analyzed (Participants) | 86
  Week 24 | -43.64 (37.606)
  Week 48: number analyzed (Participants) | 95
  Week 48 | -43.88 (36.037)
  Week 72: number analyzed (Participants) | 92
  Week 72 | -45.17 (31.571)
  Week 96: number analyzed (Participants) | 66
  Week 96 | -38.00 (52.859)
  Week 120: number analyzed (Participants) | 39
  Week 120 | -33.10 (65.888)

3. Secondary Outcome: Absolute Change in LDL-C Over Time
Description: as for outcome 1
Time Frame: Up to 120 weeks
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Overall Study Total Evinacumab
Number analyzed (Participants) | 116
mg/dL
  Week 8: number analyzed (Participants) | 109
  Week 8 | -142.1 (114.61)
  Week 24: number analyzed (Participants) | 86
  Week 24 | -132.0 (124.37)
  Week 48: number analyzed (Participants) | 95
  Week 48 | -132.8 (133.29)
  Week 72: number analyzed (Participants) | 92
  Week 72 | -135.1 (121.91)
  Week 96: number analyzed (Participants) | 66
  Week 96 | -131.4 (129.29)
  Week 120: number analyzed (Participants) | 39
  Week 120 | -132.5 (132.03)

4. Secondary Outcome: Percent Change in Apolipoprotein B (Apo B) Over Time
Description: as for outcome 1
Time Frame: Up to 120 weeks
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Overall Study Total Evinacumab
Number analyzed (Participants) | 116
Percentage of change
  Week 8: number analyzed (Participants) | 109
  Week 8 | -39.74 (25.338)
  Week 24: number analyzed (Participants) | 86
  Week 24 | -36.98 (27.574)
  Week 48: number analyzed (Participants) | 96
  Week 48 | -35.85 (29.998)
  Week 72: number analyzed (Participants) | 93
  Week 72 | -37.60 (27.292)
  Week 96: number analyzed (Participants) | 66
  Week 96 | -32.54 (39.969)
  Week 120: number analyzed (Participants) | 39
  Week 120 | -27.73 (51.722)

5. Secondary Outcome: Absolute Change in Apo B Over Time
Description: as for outcome 1
Time Frame: Up to 120 weeks
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Overall Study Total Evinacumab
Number analyzed (Participants) | 116
mg/dL
  Week 8: number analyzed (Participants) | 109
  Week 8 | -78.0 (59.78)
  Week 24: number analyzed (Participants) | 86
  Week 24 | -70.5 (61.96)
  Week 48: number analyzed (Participants) | 96
  Week 48 | -69.4 (69.95)
  Week 72: number analyzed (Participants) | 93
  Week 72 | -73.9 (61.51)
  Week 96: number analyzed (Participants) | 66
  Week 96 | -71.5 (66.66)
  Week 120: number analyzed (Participants) | 39
  Week 120 | -70.7 (76.05)

6. Secondary Outcome: Percent Change in Non-High-Density Lipoprotein Cholesterol (HDL-C) Over Time
Description: as for outcome 1
Time Frame: Up to 120 weeks
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Overall Study Total Evinacumab
Number analyzed (Participants) | 116
Percentage of change
  Week 8: number analyzed (Participants) | 109
  Week 8 | -48.47 (28.369)
  Week 24: number analyzed (Participants) | 86
  Week 24 | -46.14 (29.117)
  Week 48: number analyzed (Participants) | 95
  Week 48 | -45.15 (33.566)
  Week 72: number analyzed (Participants) | 92
  Week 72 | -46.69 (28.534)
  Week 96: number analyzed (Participants) | 66
  Week 96 | -40.88 (46.588)
  Week 120: number analyzed (Participants) | 39
  Week 120 | -35.85 (58.374)

7. Secondary Outcome: Absolute Change in Non-HDL-C Over Time
Description: as for outcome 1
Time Frame: Up to 120 weeks
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Overall Study Total Evinacumab
Number analyzed (Participants) | 116
mg/dL
  Week 8: number analyzed (Participants) | 109
  Week 8 | -153.7 (115.66)
  Week 24: number analyzed (Participants) | 86
  Week 24 | -143.9 (125.03)
  Week 48: number analyzed (Participants) | 95
  Week 48 | -144.1 (136.95)
  Week 72: number analyzed (Participants) | 92
  Week 72 | -147.3 (122.76)
  Week 96: number analyzed (Participants) | 66
  Week 96 | -144.5 (131.15)
  Week 120: number analyzed (Participants) | 39
  Week 120 | -142.9 (136.65)

8. Secondary Outcome: Percent Change in Total Cholesterol (TC) Over Time
Description: as for outcome 1
Time Frame: Up to 120 weeks
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Overall Study Total Evinacumab
Number analyzed (Participants) | 116
Percentage of change
  Week 8: number analyzed (Participants) | 109
  Week 8 | -47.04 (20.722)
  Week 24: number analyzed (Participants) | 86
  Week 24 | -44.17 (24.224)
  Week 48: number analyzed (Participants) | 95
  Week 48 | -43.78 (27.838)
  Week 72: number analyzed (Participants) | 93
  Week 72 | -44.58 (25.700)
  Week 96: number analyzed (Participants) | 66
  Week 96 | -40.33 (38.163)
  Week 120: number analyzed (Participants) | 39
  Week 120 | -36.92 (47.469)

9. Secondary Outcome: Absolute Change in TC Over Time
Description: as for outcome 1
Time Frame: Up to 120 weeks
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Overall Study Total Evinacumab
Number analyzed (Participants) | 116
mg/dL
  Week 8: number analyzed (Participants) | 109
  Week 8 | -167.3 (115.76)
  Week 24: number analyzed (Participants) | 86
  Week 24 | -157.4 (125.93)
  Week 48: number analyzed (Participants) | 95
  Week 48 | -158.2 (136.51)
  Week 72: number analyzed (Participants) | 93
  Week 72 | -160.7 (123.09)
  Week 96: number analyzed (Participants) | 66
  Week 96 | -157.2 (132.40)
  Week 120: number analyzed (Participants) | 39
  Week 120 | -153.8 (138.26)

10. Secondary Outcome: Percent Change in Triglycerides (TGs) Over Time
Description: as for outcome 1
Time Frame: Up to 120 weeks
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Overall Study Total Evinacumab
Number analyzed (Participants) | 116
Percentage of change
  Week 8: number analyzed (Participants) | 107
  Week 8 | -45.97 (26.024)
  Week 24: number analyzed (Participants) | 84
  Week 24 | -46.93 (24.582)
  Week 48: number analyzed (Participants) | 94
  Week 48 | -43.25 (37.443)
  Week 72: number analyzed (Participants) | 92
  Week 72 | -46.50 (25.826)
  Week 96: number analyzed (Participants) | 66
  Week 96 | -48.28 (24.136)
  Week 120: number analyzed (Participants) | 36
  Week 120 | -42.06 (36.945)

11. Secondary Outcome: Absolute Change in TGs Over Time
Description: as for outcome 1
Time Frame: Up to 120 weeks
Population: Here 'n' = number of evaluable participants at the specified timepoint
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Overall Study Total Evinacumab
Number analyzed (Participants) | 116
mg/dL
  Week 8: number analyzed (Participants) | 107
  Week 8 | -64.4 (89.77)
  Week 24: number analyzed (Participants) | 84
  Week 24 | -68.1 (97.29)
  Week 48: number analyzed (Participants) | 94
  Week 48 | -66.7 (97.02)
  Week 72: number analyzed (Participants) | 92
  Week 72 | -68.8 (91.52)
  Week 96: number analyzed (Participants) | 66
  Week 96 | -75.2 (107.49)
  Week 120: number analyzed (Participants) | 36
  Week 120 | -66.7 (110.95)

ADVERSE EVENTS:
Time Frame: From signing of Informed Consent to week 216
Groups:
- Overall: Includes all participants who were enrolled and received at least 1 dose or part of a dose of open-label study treatment.
Arm/Group | Overall
All-Cause Mortality (participants affected / at risk) | 2/116
Serious Adverse Events (participants affected / at risk) | 27/116
Other Adverse Events (participants affected / at risk) | 79/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=116)
Angina pectoris (Cardiac disorders) | 2 (2)
Angina unstable (Cardiac disorders) | 2 (3)
Aortic valve disease (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (2)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (2)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Supravalvular aortic stenosis (Cardiac disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1)
Chest pain (General disorders) | 2 (3)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Spinal epidural haematoma (Nervous system disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1)
Food allergy (Immune system disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Renal infarct (Renal and urinary disorders) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=116)
Nasopharyngitis (Infections and infestations) | 23 (42)
COVID-19 (Infections and infestations) | 19 (20)
Gastroenteritis (Infections and infestations) | 10 (11)
Urinary tract infection (Infections and infestations) | 10 (16)
Upper respiratory tract infection (Infections and infestations) | 9 (14)
Nausea (Gastrointestinal disorders) | 14 (17)
Diarrhoea (Gastrointestinal disorders) | 10 (21)
Abdominal pain (Gastrointestinal disorders) | 7 (10)
Toothache (Gastrointestinal disorders) | 7 (10)
Vomiting (Gastrointestinal disorders) | 7 (11)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6)
Influenza like illness (General disorders) | 17 (23)
Pyrexia (General disorders) | 10 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (20)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (10)
Headache (Nervous system disorders) | 19 (29)
Dizziness (Nervous system disorders) | 7 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (16)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Contusion (Injury, poisoning and procedural complications) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT03409744/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/44/NCT03409744/SAP_001.pdf